CLINICAL TRIAL: NCT05929586
Title: A Pragmatic Open-label, Community-based, Cluster Randomised Controlled Superiority Trial to Evaluate the Efficacy and Cost-effectiveness of Digital Data Linkage and Scheduling ('C-it') With or Without Community Data Use ('DU-it') to Increase Antenatal Clinic Uptake in Western Kenya.
Brief Title: Digital Data Linkage and Scheduling to Track Pregnancy With or Without Community Data Use to Increase Antenatal Clinic Uptake in Western Kenya.
Acronym: C-it-DU-it
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); LVCT Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-073
Record Dates: First submitted 2023-04-05; First posted 2023-07-03 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Health Systems; Electronic Community Health Information Systems; Antenatal Clinic Uptake; Pregnancy

STUDY DESIGN:
Intervention Model Description: Allocation: cluster randomised; intervention model: parallel assignment; arms: 2; allocation ratio: 1:1; restricted or stratified randomisation. Masking: none
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital data linkage and scheduling ('C-it'): The "C-it" enhanced standard of care (No Intervention): Linking facility to community digital data via linkage-app: Data between electronic Community Health Information System (eCHIS) and facility-based Kenya Electronic Medical Record (Kenya EMR) do not link. We do not have an existing digital data linkage module or app to track successful pregnancy referrals or allow the facility staff to view community contacts and vice versa. We will engage with national and county teams and software developers to build a digital data linkage module, linking eCHIS and Kenya EMR Maternal and Child Health (MCH) module.
- The combined "C-it DU-it" intervention: community data use for ANC (Experimental): Combining "C-it" and work improvement teams (WITs) for community data use: We will establish and train integrated WITs in intervention sites consisting of community health members, health facility staff and community members and train them on how they will use linkage-app. The resultant combined "C-it DU-it" intervention has three building blocks:
  We make the following assumptions about the building blocks at the bottom of figure 1.
  1. Building block 1: We assume that high-quality digital data that can trace the entire journey through pregnancy is accessible to CHVs
  2. Building block 2: We also assume that integrated work improvement teams (WITs) will have the right people around the table with clearly defined roles and responsibilities will use the data.
  3. Building block 3: Community ANC contacts will be implemented.
  Interventions: Other: The combined "C-it DU-it" intervention: community data use for ANC

INTERVENTIONS:
Other: The combined "C-it DU-it" intervention: community data use for ANC — Combining data linkage ("C-it") with work improvement teams for community data use ("DU-it") to improve antenatal clinic uptake. Our short name C-it DU-it (pronounced "see-it; do-it") is an acronym intended to convey 'seeing' linked data (C-it) and 'doing' or acting on the data (DU-it)
  Other Names: community data use (DU-it)
  Arms: The combined "C-it DU-it" intervention: community data use for ANC

SUMMARY:
The investigators propose to increase ANC uptake through a health systems strengthening approach that links digital data platforms and trains community Work Improvement Teams (WITs) to use these data to identify problems and come up with local solutions. Our short name C-it DU-it (pronounced "see-it; do-it") is an acronym intended to convey 'seeing' linked data (C-it) and 'doing' or acting on the data (DU-it). The trial design is a 2-arm, cluster-randomised controlled superiority trial in Homa Bay County to determine the efficacy of 'C-it DU-it' intervention (data use arm) to increase ANC contacts when compared to the 'C-it' enhanced standard of care (control arm).

DETAILED DESCRIPTION:
Facility and community health data is being rapidly digitised using multiple parallel systems across the 47 devolved counties in Kenya, but data do not link. Setting up community-based antenatal care (ANC) to complement facility-based ANC and data systems that link these platforms is essential to support Kenya in adopting WHO's ambitious target of 8 ANC contacts. As of February 2023, national scale up of the national electronic community health information systems (eCHIS) for standard of care is ongoing, and there are increased efforts to scale-up use of the nationally approved Kenya Electronic Medical Records (KenyaEMR) Maternal and Child Health Module (MNH) to capture ANC, delivery and postnatal (PNC) data at health facilities. Data between eCHIS and Kenya EMR do not link. There are plans within the Community Health Division at national level to link eCHIS to facility EMRs, but this has yet to be developed. The investigators propose to increase ANC uptake through a health systems strengthening approach that links digital data platforms and trains community Work Improvement Teams (WITs) to use these data to identify problems and come up with local solutions. The short name C-it DU-it (pronounced "see-it; do-it") is an acronym intended to convey 'seeing' linked data (C-it) and 'doing' or acting on the data (DU-it). The overarching research question the investigators will seek to answer is "what is the effect of 'C-it DU it' on community health systems strengthening and what is required for effective transfer and scale-up?" The investigators will use mixed methods implementation research to evaluate this in 4 counties in Western Kenya (Homa Bay, Migori, Kisumu, Kakamega) over a period of four years. The proposed methods include: (a) Realist evaluation to generate, empirically test and refine a transferrable programme theory to understand the causal relationship between context, participant response and outcomes; (b) A 2-arm, cluster-randomised controlled superiority trial in Homa Bay County to determine the efficacy of 'C-it DU-it' intervention (data use arm) to increase ANC contacts when compared to the 'C-it' enhanced standard of care (control arm); (c) Health economic evaluation and equity analysis to compare costs and catastrophic health expenditure of women accessing and engaging with ANC care and determine costs and cost-effectiveness of C-it Du-it from a health systems perspective; and (d) Qualitative interviews will assess transferability and iterative scale-up of C-it DU-it across the three remaining counties using toolkits developed in Homa Bay. This protocol describes the pragmatic cluster randomised trial and health economic evaluation. The realist evaluation and scale up will be addressed in a separate sister protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of all ages willing to participate
* Written informed consent
* A resident of the study area (catchment area) for the duration of the pregnancy
* Delivered and still within the 6-week post-partum period.

Exclusion Criteria:

* Currently enrolled in another interventional study targeting pregnant women
* Outside the 6-week post-partum period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 1440 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Increasing antenatal clinic uptake | 14 months
  The proportion of women having at least eight ANC contacts during the antenatal period, defined as either a scheduled ANC visit in the facility or a scheduled ANC contact with a CHV in the community assessed at birth (or within the first 6-8 weeks for home births) using the ANC cards.
Estimate socioeconomic impact and access to social protection | 14 months
  Defined as the proportion of women using financial coping strategies and their frequency and distribution
Estimate the costs to pregnant women and their households | 14 months
  Absolute costs to the pregnant woman and their household and the costs as a proportion of the pregnant woman and their household's monthly income or expenditure/consumption will be calculated for the following variables:
  * Out-of-pocket medical costs
  * Out-of-pocket non-medical costs
  * Lost income, time, and productivity

SECONDARY OUTCOMES:
The proportion of women having at least four scheduled ANC visits in the facility | 14 months
  assessed at birth (or within the first 6-8 weeks after birth for home births) using the ANC cards.
The proportion of women having at least eight scheduled ANC visits in the facility | 14 months
  assessed at birth (or within the first 6-8 weeks after birth for home births) using the ANC cards.
The frequency (count) of scheduled ANC visits | 14 months
  assessed at birth (or within the first 6-8 weeks after birth for home births) using the ANC cards.
The frequency (count) of of ANC visits in the community | 14 months
  assessed at birth (or within the first 6-8 weeks after birth for home births) using the ANC cards.
Early antenatal clinic attendance | 14 months
  The proportion of women with a first ANC contact before 16 weeks gestation.
Quality of antenatal care | 14 months
  * The proportion of women with at least three courses of IPTp
  * The proportion of women who received iron and folate for 90 days.
  * The proportion of women receiving testing and management for HIV.
  * The proportion of women receiving testing and management for malaria.
  * The proportion of women receiving testing and management for syphilis.
  * The proportion of women receiving testing and management for anaemia.
Uptake of skilled birth attendance. | 14 months
  The proportion of women who had a skilled birth attendance.
Reducing the risk of adverse pregnancy outcomes. | 14 months
  The proportion of women with adverse pregnancy outcomes- defined as a composite of foetal loss (stillbirth or spontaneous miscarriage), low birth weight or neonatal mortality)
prevalence of catastrophic health expenditure (CHE) of accessing ANC care with "C-it" enhanced standard of care | 14 months
  CHE prevalence at two World Health Organization-defined thresholds: out-of-pocket medical costs of more than 10% of a patient household's total monthly expenditure/consumption (10%-threshold); and out-of-pocket medical costs of more than 40% of a patient household's monthly capacity to pay (non-food/housing/utilities expenditure/consumption)
  • A sensitivity analysis of the proportion of women's households incurring CHE due to pregnancy and ANC visits using varying additional recognised calculations and thresholds including, as per WHO Tuberculosis Patient Cost Survey methodology, the addition of non-medical out-of-pocket costs and lost income in the numerator
Cost-effectiveness of "C-it" and "C-it DU-it" intervention | 14 months
  Incremental cost-effectiveness ratios (ICERs) compared across trial arms
Assess equity of access to ANC and "C-it" and "C-it DU-it" intervention. | 14 months
  Equity of access to ANC and the interventions will be evaluated by exploratory distributional (or "extended") cost-effectiveness analysis of the intervention across the following sub-groups: poverty quintiles, age groups including adolescents vs adults, study sites, HIV status, and by eligibility for health insurance including NHIF and Linda Mama.

OTHER OUTCOMES:
Improving uptake of four ANC tests. | 14 months
  The proportion of women receiving testing and management of all four common conditions in pregnancy (HIV, syphilis, malaria, anaemia).
Improving uptake of HIV prevention services. | 14 months
  The proportion of HIV-negative women receiving testing and management for HIV in the 3rd trimester or at delivery.
  The proportion of HIV-exposed infants with negative HIV PCR DNA tests at 6-8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Taegtmeyer, PhD, Principal Investigator — Liverpool School of Tropical Medicine; Tom Wingfield, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- KEMRI Centre for Global Health Research, Homa Bay, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via data transfer agreements with the collaborating institutions to minimise the risk of unauthorised analysis beyond the scope of the agreed parameters. The full protocol will be available on request to any interested professional and may be published in a peer-reviewed journal or deposited in an online repository. Individual, de-identified participant data will be made available for meta-analyses as soon as the data analysis is completed, with the understanding that the meta-analysis results will not be published before the individual trial results without the prior agreement of the investigators. The de-identified data set of the complete participant-level data will be available for sharing purposes. A Data Access Committee will consider all requests for data for secondary analysis to ensure that the use of data is within the terms of consent and ethics approval and in line with the Kenya Data Protection Act 2019.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The full anonymised research database will be made publicly available as soon as the full study findings have been published or based on any data requests that may occur during the study or analysis is still ongoing.
Access Criteria: Data access will be provided to researchers after a proposal has been approved by an independent review committee identified for this purpose. An agreement on how to collaborate will be reached based on any overlap between the proposal and any ongoing efforts. Proposals can be directed to email addresses provided in the publications and websites. To gain access, data requesters will need to sign a data-sharing agreement.